CLINICAL TRIAL: NCT01673841
Title: Relation Between Mixed Venous Oxygen Saturation and Cerebral Oxygen Saturation Measured by Absolute and Relative Near-infrared Spectroscopy During Off-pump Coronary Artery Bypass Grafting.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgian Foundation for Cardiac Surgery (Unknown); CAS Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2009/126
Record Dates: First submitted 2012-08-17; First posted 2012-08-28 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Elective Off-pump Coronary Artery Bypass Grafting
Keywords: bypass grafting
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relative + absolute cerebral oxygen saturation.
  Interventions: Procedure: Relative and absolute cerebral oxygen saturation (rScO2) measurements.

INTERVENTIONS:
Procedure: Relative and absolute cerebral oxygen saturation (rScO2) measurements.

SUMMARY:
In this clinical study the investigators compared mixed venous oxygen saturation (SmvO2) with relative and absolute cerebral oxygen saturation (rScO2) measurements. They hypothesized that previously reported contradictory results regarding the equivalence of SmvO2 and rScO2 might be related to time delay issues and to the measurement technology.

42 consenting patients undergoing elective off-pump coronary artery bypass grafting were included. 4 disposable oxygenation sensors were applied bilaterally on the patient's forehead for continuous, non-invasive registration of rScO2. The sensors of one monitor were placed just above the eyebrows, and the sensors of the other monitor were placed just above the former sensors. The sensors placement was determined at random by a computerized randomization list. SmvO2 was measured continuously via a pulmonary artery catheter. All variables were recorded continuously. The study ended at the end of the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective off-pump coronary artery bypass grafting for at least 3-vessel coronary artery disease were eligible.

Exclusion Criteria:

* Patients with arteriovenous shunts, intracardiac shunts, a previous history of cerebrovascular accident, or stenosis of the internal carotid artery of > 60% were excluded.

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective off-pump coronary artery bypass grafting.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Correlation and time delay between mixed venous and cerebral oxygen saturation during off-pump coronary artery bypass grafting. | 4 hours during an operation of average 5 hours (during off-pump coronary artery bypass grafting).
  Mixed venous oxygen saturation was measured continuously via a pulmonary artery catheter. Cerebral oxygen saturation was measured with near-infrared spectroscopy; the INVOS monitor to obtain relative measurements, and the Foresight monitor to obtain absolute data.

SECONDARY OUTCOMES:
The response of cerebral oxygen saturation to major haemodynamic disturbances. | 2 hours after start of operation (during placement of deep pericardial stitches).
  Percentage difference between the cerebral oxygen saturation value just before heart retraction and the value at the different time moments.

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Moerman, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be